CLINICAL TRIAL: NCT01175382
Title: Combined Behavioral and Drug Treatment of Overactive Bladder in Men
Acronym: COBALT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Kathryn Burgio, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DK082548-01A1 (NIH)
Record Dates: First submitted 2010-08-03; First posted 2010-08-04 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-04

CONDITIONS: Overactive Bladder; Lower Urinary Tract Symptoms
Keywords: Male Urogenital Diseases; Urinary Bladder, overactive; Behavioral Medicine; Drug Therapy
MeSH Terms: conditions — Urinary Bladder, Overactive; Lower Urinary Tract Symptoms; Male Urogenital Diseases | interventions — Tolterodine Tartrate; Tamsulosin; Drug Therapy

STUDY DESIGN:
Intervention Model Description: The design of this study is a 3 group randomized trial. Group 1 was randomized to drug only for the first 6 weeks, followed by a step up to drug plus behavior from 6 weeks to 12 weeks. Group 2 was randomized to behavior only for the first 6 weeks, followed by a step up to behavior plus drug from 6 weeks to 12 weeks. Group 3 was randomized to behavior plus drug from baseline to 12 weeks.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Behavioral Treatment alone (Active Comparator): Behavioral treatment is implemented in 4 clinic visits over a period of 6 weeks, followed by 6 weeks of combined behavioral + drug therapy. Behavioral treatment consists of behavioral training and includes skills and strategies for postponing urination, controlling urgency and preventing urge incontinence. This includes pelvic floor muscle training, incremental delayed voiding, and daily bladder diaries, supplemented with instructions for daily home practice between clinic visits. In addition to daytime training, nocturia is managed with fluid restriction (3 hours before bedtime and during the night) and with urge strategies.
  Interventions: Behavioral: Behavioral training
- Drug Therapy (Tolterodine + tamsulosin) (Active Comparator): Drug therapy for 6 weeks implemented in a clinic visit with telephone follow-up at 3 weeks, followed by 6 weeks of combined drug + behavioral therapy. Participants in the drug group will receive an anti-muscarinic (sustained release tolterodine 4 mg) + an alpha blocker (tamsulosin 0.4mg daily).
  Interventions: Drug: Tolterodine + tamsulosin
- Combined Behavioral + Drug Therapy (Experimental): Combined behavioral and drug therapy implemented in 4 clinic visits over a period of 6 weeks, followed by an additional 6 weeks of combined therapy. Behavioral treatment consists of behavioral training and includes skills and strategies for postponing urination, controlling urgency and preventing urge incontinence. This includes pelvic floor muscle training, incremental delayed voiding, and bladder diaries, supplemented with instructions for daily home practice. Nocturia is managed with fluid restriction (3 hours before bedtime and during the night) and with urge strategies. Drug therapy consists of an anti-muscarinic (sustained release tolterodine 4 mg) + an alpha blocker (tamsulosin 0.4mg daily).
  Interventions: Other: Combined Behavioral + Drug Therapy

INTERVENTIONS:
Behavioral: Behavioral training — Behavioral treatment consists of skills and strategies for postponing urination, controlling urgency and preventing urge incontinence. This includes pelvic floor muscle training, urge suppression techniques, delayed voiding, and daily bladder diaries to track increasing voiding intervals and enhance awareness of bladder habits. Training is supplemented with instructions for daily home practice between clinic visits. In addition to daytime training, nocturia is managed with fluid restriction (3 hours before bedtime and during the night) and with urge strategies.
  Other Names: Urge suppression; Delayed voiding; Pelvic floor muscle training
  Arms: Behavioral Treatment alone
Drug: Tolterodine + tamsulosin — Patients in drug therapy receive an anti-muscarinic (long acting tolterodine 4 mg daily) and an alpha blocker (tamsulosin 0.4 mg daily).
  Other Names: Flomax; Detrol Long-Acting (LA); Tolterodine tartrate
  Arms: Drug Therapy (Tolterodine + tamsulosin)
Other: Combined Behavioral + Drug Therapy — Combined behavioral and drug therapy implemented in 4 clinic visits over a period of 6 weeks, followed by an additional 6 weeks of combined therapy. Behavioral treatment consists of behavioral training and includes skills and strategies for postponing urination, controlling urgency and preventing urge incontinence. This includes pelvic floor muscle training, incremental delayed voiding, and bladder diaries, supplemented with instructions for daily home practice. Nocturia is managed with fluid restriction (3 hours before bedtime and during the night) and with urge strategies. Drug therapy consists of an anti-muscarinic (sustained release tolterodine 4 mg) + an alpha blocker (tamsulosin 0.4mg daily).
  Arms: Combined Behavioral + Drug Therapy

SUMMARY:
The primary aim of this project is to evaluate the effectiveness of combined behavioral + drug therapy compared to behavioral treatment alone and drug therapy alone as a way to improve outcomes in the treatment of OAB symptoms in men. We hypothesize that combined therapy will result in better outcomes than either behavioral or drug therapy alone. The second aim is to compare two methods of implementing combined therapy: simultaneously as initial therapy vs. stepped therapy, in which therapies are combined following initial behavioral or drug therapy alone. The third aim is to examine the costs and cost-effectiveness of combined behavioral + drug therapy compared to behavioral or drug therapy alone.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a very common, distressing condition that manifests as bothersome symptoms of urgency, frequent urination, urge incontinence, and nocturia, and impacts the lives of millions of men. OAB symptoms are most often treated with pharmacologic therapies (alpha-blocking agents and/or antimuscarinic agents) or behavioral treatments. Although drug therapies (even combined drug therapies) and behavioral treatments reduce OAB symptoms, few patients are completely cured with either treatment alone. Therefore, there is a need to improve interventions for this common problem. The primary purpose of this study is to test the effectiveness of combining behavioral treatment and drug therapy as a way to improve outcomes in the treatment of OAB symptoms in men. This is a 3-site, 2-stage, 3-arm randomized clinical trial of behavioral treatment, drug therapy, and combined drug + behavioral therapy for men with OAB, to examine the efficacy of combined therapy and whether it yields higher success rates than either therapy alone. 204 men with OAB were enrolled and randomized to 1) drug therapy alone followed by combined therapy, 2) behavioral treatment alone followed by combined therapy, or 3) combined therapy as initial treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling men
2. Age 40 years or older
3. Patient-reported urgency and 9.0 or more voids per 24-hour day (on average) on the 7-day baseline bladder diary.

Exclusion Criteria:

1. Urinary flow rate < 8.0 mL/sec on a void greater than 125 ml.
2. Post-void residual volume greater than 150 mL (based on bladder ultrasound after voiding in the presence of a normal urge to urinate).
3. Urinary tract infection (defined as growth of greater than 10,000 colonies per ml of a urinary pathogen on urine culture). Patients will be referred for treatment with antibiotics and may be enrolled if OAB symptoms persist after the infection is resolved.
4. Transurethral resection of the prostate (TURP), simple prostatectomy, or other benign prostatic hypertrophy (BPH) related surgery within the past 5 years.
5. Current active treatment for prostate cancer.
6. History of radical prostatectomy.
7. Previous artificial urinary sphincter, sling procedure, bladder-injection of botulinum toxin, or implanted sacral neuromodulation device.
8. Poorly controlled diabetes (glycosylated hemoglobin >9.0 within last 3 months). Subjects with poorly controlled diabetes will be offered enrollment if the OAB symptoms persist after the diabetes is controlled appropriately.
9. Hematuria on microscopic examination in the absence of infection. A urologic consultation will be recommended and enrollment will depend on clearance by a urologist and agreement by the Site PI that entry into the treatment protocol is not contraindicated.
10. Any unstable medical condition (particularly: cancers under active treatment, decompensated congestive heart failure, history of malignant arrhythmias, unstable angina, diagnosed by history or physical exam).
11. Neurologic conditions such as Parkinson's, spinal cord injury, multiple sclerosis, or myasthenia gravis.
12. Impaired mental status. Patients who screen as probable dementia on the Mini-Cog.
13. Contraindications to the study drugs (tolterodine and tamsulosin) including history of postural hypotension with syncope, history of acute urinary retention requiring catheterization, narrow angle glaucoma, or history of gastric retention.
14. Hypersensitivity to tolterodine or tamsulosin.
15. Current use of an alpha blocker agent. Evaluation will be delayed until the drug has been discontinued for 2 weeks.
16. Current use of an anti-muscarinic agent for OAB. Evaluation will be delayed until the drug has been discontinued for 2 weeks.
17. If on a diuretic, dose has not been stable for at least 4 weeks.
18. If taking dutasteride or finasteride, dose has not been stable for at least 6 months.
19. If on an antibiotic for prostatitis. Patients will be offered re-evaluation if OAB symptoms persist when antibiotics are completed.
20. Full course of behavioral training.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2010-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn L Burgio, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Emory University, Atlanta, Georgia
  - University of Texas Health Science Center San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Funada S, Yoshioka T, Luo Y, Sato A, Akamatsu S, Watanabe N. Bladder training for treating overactive bladder in adults. Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD013571. doi: 10.1002/14651858.CD013571.pub2. PMID 37811598
- [Derived] Burgio KL, Kraus SR, Johnson TM 2nd, Markland AD, Vaughan CP, Li P, Redden DT, Goode PS. Effectiveness of Combined Behavioral and Drug Therapy for Overactive Bladder Symptoms in Men: A Randomized Clinical Trial. JAMA Intern Med. 2020 Mar 1;180(3):411-419. doi: 10.1001/jamainternmed.2019.6398. PMID 31930360

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual: July 2010, Primary Completion Date: July 2015 and Study Completion Date: July 2015. Recruitment location: University of Alabama at Birmingham.
Pre-assignment Details: Sample sizes reported for analysis differs from the sample size in the Participant Flow Module for outcomes in patient satisfaction, perception of improvement and bothersome side effects due to patients, either not completing the form, or non-response to the questions, although they still enrolled in the study (applies for both 6 &12 week analysis)
Groups:
- Behavioral Treatment Alone: Behavioral treatment implemented in 4 clinic visits over a period of 6 weeks, followed by 6 weeks of combined behavioral + drug therapy. Behavioral treatment consists of skills and strategies for postponing urination, controlling urgency, and preventing urge incontinence. This includes pelvic floor muscle training, urge suppression techniques, incremental delayed voiding, and daily bladder diaries to track increasing voiding intervals and enhance awareness of bladder habits. Training is supplemented with instructions for daily home practice between clinic visits. In addition to daytime training, nocturia is managed with fluid restriction (3 hours before bedtime and during the night) and with urge strategies.
- Drug Therapy Alone: Drug therapy for 6 weeks implemented in a clinic visit with telephone follow-up at 3 weeks, followed by 6 weeks of combined drug + behavioral therapy. Participants receive an anti-muscarinic (sustained release tolterodine 4 mg) + an alpha blocker (tamsulosin 0.4mg daily).
- Combined Behavioral + Drug Therapy: Combined behavioral and drug therapy implemented in 4 clinic visits over a period of 6 weeks, followed by an additional 6 weeks of combined therapy. Behavioral treatment consists of skills and strategies for postponing urination, controlling urgency and preventing urge incontinence. This includes pelvic floor muscle training, urge suppression techniques, incremental delayed voiding, and bladder diaries to track increasing voiding intervals and enhance awareness of bladder habits. Training is supplemented with instructions for daily home practice between clinic visits. In addition to daytime training, nocturia is managed with fluid restriction (3 hours before bedtime and during the night) and with urge strategies. Drug therapy consists of an anti-muscarinic (sustained release tolterodine 4 mg) + an alpha blocker (tamsulosin 0.4mg daily).
Period: Overall Study
Arm/Group | Behavioral Treatment Alone | Drug Therapy Alone | Combined Behavioral + Drug Therapy
Started | 71 | 68 | 65
Completed | 63 | 61 | 59
Not Completed | 8 | 7 | 6
Not completed — Lost to Follow-up | 4 | 3 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — No longer having problem | 1 | 0 | 1
Not completed — Unable/unwilling to attend visits | 3 | 1 | 2
Not completed — Unwilling to follow protocol | 0 | 1 | 0
Not completed — Unable to tolerate study meds | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Treatment Alone | Drug Therapy Alone | Combined Behavioral + Drug Therapy | Total
Number analyzed (Participants) | 71 | 68 | 65 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (10.9) | 65.5 (11.0) | 63.2 (11.6) | 64.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 71 | 68 | 65 | 204
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 14 | 20 | 20 | 54
  Other | 9 | 4 | 4 | 17
  White | 48 | 44 | 41 | 133
Marital Status [Number; unit: participants]
  Single | 13 | 15 | 16 | 44
  Married | 40 | 34 | 41 | 115
  Divorced | 16 | 15 | 7 | 38
  Widowed | 2 | 4 | 1 | 7
Living Status [Number; unit: participants]
  Alone | 14 | 19 | 13 | 46
  With Someone | 51 | 43 | 45 | 139
  Other | 6 | 6 | 7 | 19
Earned Wages Outside Home [Number; unit: participants]
  Yes | 28 | 28 | 30 | 86
  No | 43 | 40 | 35 | 118

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Urination After 6-week Intervention (Last Observation Carried Forward)
Description: Bladder diaries completed by subjects prior to randomization and following the first phase of treatment was used to calculate changes in frequency of urination.
Time Frame: From Baseline to 6 Weeks
Measure: Mean (Standard Deviation); unit: voids per day
Groups:
- Behavioral Treatment Alone: Behavioral treatment consists of behavioral training and includes skills and strategies for postponing urination, controlling urgency and preventing urge incontinence. This includes pelvic floor muscle training, incremental delayed voiding, and bladder diaries, supplemented with instructions for daily home practice.
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
voids per day | 2.7 (2.4) | 1.5 (2.3) | 3.3 (2.2)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance used to compare mean changes from baseline to 6 weeks among groups adjusting for baseline values and age. Last Observation Carried Forward was used for imputation of missing data; Test type: Superiority or Other; p < .0001, ANOVA

2. Primary Outcome: Change in Frequency of Urination From 6 Weeks to 12 Weeks (Last Observation Carried Forward)
Description: Bladder diaries completed by subjects prior to randomization and following each phase of treatment were used to calculate changes in frequency of urination.
Time Frame: Change from 6 weeks to 12 weeks
Measure: Mean (Standard Deviation); unit: Voids per day
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
Voids per day | 0.7 (1.2) | 1.4 (1.9) | 0.2 (1.0)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance to test for differences in mean change from 6 weeks to 12 weeks in voiding frequency controlling for age and 6 week frequency. Last Observation Carried Forward was used to impute missing data; Test type: Superiority or Other; p = .0013, ANCOVA

3. Primary Outcome: Change in Frequency of Urination From Baseline to 12 Weeks (Last Observation Carried Forward)
Description: Bladder diaries completed by subjects prior to randomization and following the second phase of treatment were used to calculate changes in frequency of urination
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Voids per day
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
Voids per day | 3.3 (2.5) | 2.9 (2.5) | 3.5 (2.3)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance testing whether mean change in 24-hour voiding frequency differed among the groups after adjusting for baseline voiding frequency and age. Last Observation Carried Forward was used to impute missing data; Test type: Superiority or Other; p = 0.2933, ANCOVA

4. Secondary Outcome: Change in Urgency From Baseline to 6 Weeks (Last Observation Carried Forward)
Description: Bladder diaries completed prior to randomization and following each phase of treatment will be used to calculate changes in urgency associated with each void and incontinent episode using the Indevus Urgency Severity Scale (IUSS). IUSS asks patients about the degree of urgency, as meant to describe the urge to urinate. Patients are asked to rate the degree of urgency and its impact on the completion of activity or tasks during the time that the urgency sensation is present and before reaching the toilet for a toilet void. Four distinct, subjective degrees of urgency severity were identified, including 1) no sensation of urgency, 2) awareness of urgency but easily tolerated, 3) urgency that is somewhat uncomfortable and 4) extreme urgency discomfort.
Time Frame: From Baseline to 6 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
units on a scale | -0.1 (0.5) | 0.1 (0.5) | 0.2 (0.6)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance used to test means changes among the groups adjusting for baseline values and age. Last Observation Carried Forward was used to impute missing data; Test type: Superiority or Other; p = 0.0051, ANCOVA

5. Secondary Outcome: Change in Urinary Incontinence From Baseline to 6 Weeks (Last Observation Carried Forward)
Description: Bladder diaries completed prior to randomization and following each phase of treatment will be used to calculate changes in frequency of incontinence episodes.
Time Frame: From Baseline to 6 Weeks
Measure: Mean (Standard Deviation); unit: episodes per week
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
episodes per week | 3.4 (7.0) | 3.1 (10.6) | 5.2 (8.7)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance comparing mean change score among groups controlling for age and baseline score; Test type: Superiority or Other; p = .1402, ANCOVA

6. Secondary Outcome: Change in Nocturia From Baseline to 6 Weeks (Last Observation Carried Forward)
Description: Bladder diaries completed prior to randomization and following each phase of treatment will be used to calculate changes in frequency of nocturia.
Time Frame: From Baseline to 6 Weeks
Measure: Mean (Standard Deviation); unit: voids per night
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
voids per night | 0.7 (1.0) | 0.4 (0.9) | 0.8 (1.1)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance comparing mean change in Nocturia among groups adjusting for baseline values of nocturia and age. Last Observation Carried Forward was used to impute missing data; Test type: Superiority or Other; p = 0.0015, ANCOVA

7. Secondary Outcome: Change in Overactive Bladder Questionnaire (OAB-q) From Baseline to 6 Weeks (Last Observation Carried Forward)
Description: Change from baseline on the OAB-q to measure symptom bother and condition-specific health-related quality of life. This questionnaire asks about how much you have been bothered by selected bladder symptoms during the past 4 weeks. Scale ranges from 8 to 48 with higher scores indicating a greater degree of bother.
Time Frame: From Baseline to 6 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
units on a scale | 19.9 (20.8) | 20.2 (27.5) | 37.5 (31.8)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance comparing mean change in Overactive Bladder Questionnaire from baseline to 6 weeks among groups after controlling for baseline value and age. Last Observation Carried Forward was used to impute missing data; Test type: Superiority or Other; p < .0001, ANCOVA

8. Secondary Outcome: Change in International Prostate Symptom Score (I-PSS) From Baseline to 6 Weeks. (Last Observation Carried Forward)
Description: Change from baseline to 6 weeks on the International Prostate Symptom Score (IPSS) to measure urinary symptoms related to benign prostatic hypertrophy (BPH). The I-PSS is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
Time Frame: From Baseline to 6 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
units on a scale | 4.0 (3.9) | 4.4 (5.9) | 7.9 (5.2)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance comparing mean chance in IPSS from baseline to 6 weeks among groups controlling for baseline IPSS values and age. Last Observation Carried Forward was used to impute missing data; Test type: Superiority or Other; p < .0001, ANCOVA

9. Secondary Outcome: Patient Satisfaction
Description: Patient global ratings of satisfaction using the validated Patient Satisfaction Question
Time Frame: From Baseline to 6 Weeks
Population: Sample sizes reported for analysis differs from the sample size in the Participant Flow Module for Outcomes in patient satisfaction, perception of improvement and bothersome side effects due to patients, either not completing the form or non-response to the questions, although they still enrolled in the study (applies for both 6 &12 week analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 64 | 65 | 61
Participants
  Much Better | 13 | 9 | 24
  Better | 39 | 33 | 31
  About the Same | 12 | 22 | 6
  Worse | 0 | 1 | 0
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Test type: Superiority or Other; p = 0.0022, Cochran-Mantel-Haenszel

10. Secondary Outcome: Patient Perceptions of Improvement
Description: Patient global ratings of improvement using the validated Estimated Percent Improvement and Global Perception of Improvement
Time Frame: From Baseline to 6 Weeks
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 64 | 65 | 61
Participants
  Completely | 18 | 13 | 30
  Somewhat Satisfied | 42 | 41 | 30
  Somewhat Dissatisfied | 3 | 8 | 1
  Very Dissatified | 1 | 3 | 0
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Test type: Superiority or Other; p = .0222, Cochran-Mantel-Haenszel

11. Secondary Outcome: How Bothersome Were Side Effects? 6 Week Report
Description: Ordinal Rating regarding how bothersome side effects were
Time Frame: From Baseline to 6 weeks
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 64 | 65 | 61
Participants
  No Side effects | 33 | 12 | 8
  Not at all bothersome | 22 | 9 | 13
  A little | 6 | 20 | 29
  Somewhat | 3 | 18 | 10
  Extremely | 0 | 6 | 1
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Test type: Superiority or Other; p = .0217, Cochran-Mantel-Haenszel

12. Secondary Outcome: Change in Urgency Score From 6 Weeks to 12 Weeks (Last Observation Carried Forward)
Description: Bladder diaries completed by subjects prior to randomization and following each phase of treatment will be used to calculate changes in urgency associated with each void and incontinent episode using the Indevus Urgency Severity Scale (IUSS). IUSS asks patients about the degree of urgency, as meant to describe the urge to urinate. Patients are asked to rate the degree of urgency and its impact on the completion of activity or tasks during the time that the urgency sensation is present and before reaching the toilet for a toilet void. Four distinct, subjective degrees of urgency severity were identified, including 1) no sensation of urgency, 2) awareness of urgency but easily tolerated, 3) urgency that is somewhat uncomfortable and 4) extreme urgency discomfort.
Time Frame: Change from 6 weeks to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
units on a scale | 0.1 (0.4) | 0.1 (0.4) | 0.1 (0.4)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance used to test whether mean changes in Urgency Score from 6 weeks to 12 weeks differed among groups after controlling for age and 6 week Urgency Score. Last Observation Carried Forward was used to impute missing values; Test type: Superiority or Other; p = 0.6690, ANCOVA

13. Secondary Outcome: Change in Urinary Incontinence From 6 Weeks to 12 Weeks (Last Observation Carried Forward)
Description: Bladder diaries completed by subjects prior to randomization and following each phase of treatment will be used to calculate changes in frequency of incontinence episodes.
Time Frame: Change from 6 weeks to 12 weeks
Measure: Mean (Standard Deviation); unit: Episodes per week
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
Episodes per week | 1.3 (3.6) | 1.5 (4.5) | 0.0 (2.7)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance to test whether mean change in Incontinence Episodes from 6 weeks to 12 weeks differed among groups after controlling for age and frequency of incontinence episodes at 6 weeks. Last Observation Carried Forward was used to impute missing values; Test type: Superiority or Other; p = 0.0812, ANCOVA

14. Secondary Outcome: Change in Nocturia From 6 Weeks to 12 Weeks (Last Observation Carried Forward)
Description: Bladder diaries completed by subjects prior to randomization and following each phase of treatment will be used to calculate changes in frequency of nocturia
Time Frame: Change from 6 weeks to 12 weeks
Measure: Mean (Standard Deviation); unit: Voids per night
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
Voids per night | 0.1 (0.6) | 0.3 (0.9) | 0.1 (0.6)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance used to test whether mean changes in nocturia from 6 weeks to 12 weeks differed among groups after controlling for age and 6 week nocturia frequency. Last Observation Carried Forward was used to impute missing values; Test type: Superiority or Other; p = 0.5578, ANCOVA

15. Secondary Outcome: Change in Overactive Bladder Questionnaire (OAB-q) From 6 to 12 Weeks (Last Observation Carried Forward)
Description: Change from 6 weeks to 12 weeks on the OAB-q to measure symptom bother and condition-specific health-related quality of life. This questionnaire asks about how much you have been bothered by selected bladder symptoms during the past 4 weeks. Scale ranges from 8 to 48 with higher scores indicating a greater degree of bother.
Time Frame: Change from 6 week to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
units on a scale | 17.3 (20.9) | 10.8 (17.9) | 4.6 (13.9)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance to test whether mean change in Overactive Bladder Questionnaire (OAB-q) from 6 to 12 weeks differed among groups after controlling for age and 6 week OAB-q score. Last Observation Carried Forward was used to impute missing values; Test type: Superiority or Other; p = 0.0279, ANCOVA

16. Secondary Outcome: Change in International Prostate Symptom Score (IPSS) From 6 to 12 Weeks (Last Observation Carried Forward)
Description: Change from 6 weeks to 12 weeks on the International Prostate Symptom Score (IPSS) to measure urinary symptoms related to BPH.The I-PSS is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
Time Frame: Change from 6 weeks to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
units on a scale | 2.7 (4.4) | 2.2 (4.0) | 0.8 (3.0)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance to test whether mean change in the International Prostate Symptom Scale (IPSS) from 6 to 12 weeks differed among groups; Test type: Superiority or Other; p = 0.2553, ANCOVA

17. Secondary Outcome: Patient Perception of Improvement at 12 Weeks
Description: as for outcome 10
Time Frame: 12 weeks post randomization
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 62 | 61 | 59
Participants
  Much Better | 28 | 26 | 30
  Better | 27 | 26 | 26
  About the Same | 5 | 9 | 3
  Worse | 2 | 0 | 0
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Test type: Superiority or Other; p = 0.3165, Cochran-Mantel-Haenszel

18. Secondary Outcome: Satisfaction With Progress at 12 Weeks
Description: Patient global ratings of satisfaction using the validated Patient Satisfaction Question.
Time Frame: 12 weeks post randomization
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 62 | 61 | 59
Participants
  Completely | 32 | 32 | 28
  Somewhat Satisfied | 26 | 28 | 29
  Somewhat Dissatisfied | 3 | 0 | 1
  Very Dissatisfied | 1 | 1 | 1
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Test type: Superiority or Other; p = 0.8153, Cochran-Mantel-Haenszel

19. Secondary Outcome: How Bothersome Were Side Effects? 12 Week Report
Description: Ordinal Rating regarding how bothersome side effects were
Time Frame: 12 weeks post randomization
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 62 | 61 | 59
Participants
  No Side Effect | 13 | 9 | 12
  Not at all bothersome | 17 | 12 | 10
  A little | 16 | 27 | 16
  Somewhat | 14 | 12 | 19
  Extremely | 2 | 1 | 2
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Test type: Superiority or Other; p = 0.5536, Cochran-Mantel-Haenszel

20. Secondary Outcome: Change in Nocturia Measured From Baseline to 12 Weeks (Last Observation Carried Forward)
Description: Bladder diaries completed by subjects prior to randomization and following each phase of treatment will be used to calculate changes in the frequency nocturia
Time Frame: From Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: voids per night
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
voids per night | 0.8 (1.0) | 0.7 (1.0) | 0.9 (1.0)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance testing whether mean change in Nocturia frequency differed among the groups after adjusting for baseline Nocturia frequency and age. Last Observation Carried Forward was used to impute missing data; Test type: Superiority or Other; p = 0.2035, ANCOVA

21. Secondary Outcome: Change in Urgency Score From Baseline to 12 Weeks (Last Observation Carried Forward)
Description: Bladder diaries completed by subjects prior to randomization and following each phase of treatment will be used to calculate changes in frequency of urgency associated with each void and incontinent episode using the Indevus Urgency Severity Scale (IUSS). IUSS asks patients about the degree of urgency, as meant to describe the urge to urinate. Patients are asked to rate the degree of urgency and its impact on the completion of activity or tasks during the time that the urgency sensation is present and before reaching the toilet for a toilet void. Four distinct, subjective degrees of urgency severity were identified, including 1) no sensation of urgency, 2) awareness of urgency but easily tolerated, 3) urgency that is somewhat uncomfortable and 4) extreme urgency discomfort.
Time Frame: From Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
units on a scale | 0.0 (0.5) | 0.1 (0.6) | 0.2 (0.6)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance testing whether mean change in Urgency Score differed among the groups after adjusting for Urgency Scoe and age. Last Observation Carried Forward was used to impute missing data; Test type: Superiority or Other; p = .0549, ANCOVA

22. Secondary Outcome: Change in Urinary Incontinence Episodes From Baseline to 12 Weeks (Last Observation Carried Forward)
Description: Bladder diaries completed by subjects prior to randomization and following each phase of treatment will be used to calculate changes in frequency of urination
Time Frame: From Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: voids per day
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
voids per day | 4.6 (8.5) | 4.6 (10.1) | 5.2 (8.4)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance testing whether mean change in Incontinent Episodes differed among the groups after adjusting for baseline Incontinent episodes frequency and age. Last Observation Carried Forward was used to impute missing data; Test type: Superiority or Other; p = 0.5070, ANCOVA

23. Secondary Outcome: Change in Overactive Bladder Questionnaire (OAB-q) From Baseline to 12 Weeks (Last Observation Carried Forward)
Description: Change from baseline to 12 weeks on the OAB-q to measure symptom bother and condition-specific health-related quality of life. This questionnaire asks about how much you have been bothered by selected bladder symptoms during the past 4 weeks. Scale ranges from 8 to 48 with higher scores indicating a greater degree of bother.
Time Frame: From Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
units on a scale | 37.3 (31.8) | 31.0 (29.8) | 42.1 (34.1)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance testing whether mean change in Overactive Bladder Questionnaire differed among the groups after adjusting for baseline Overactive Bladder Questionnaire Score and age. Last Observation Carried Forward was used to impute missing data; Test type: Superiority or Other; p = .0529, ANCOVA

24. Secondary Outcome: Change in International Prostate Symptom Score (I-PSS) From Baseline to 12 Weeks (Last Observation Carried Forward)
Description: Change from Baseline to 12 weeks on the International Prostate Symptom Score (I-PSS) to measure urinary symptoms related to BPH. The I-PSS is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
Time Frame: From Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Treatment Alone | Drug Therapy (Tolterodine + Tamsulosin) | Combined Behavioral + Drug Therapy
Number analyzed (Participants) | 71 | 68 | 65
units on a scale | 6.7 (5.5) | 6.7 (6.2) | 8.8 (5.7)
Statistical Analysis 1: Comparison: Behavioral Treatment Alone vs Drug Therapy (Tolterodine + Tamsulosin) vs Combined Behavioral + Drug Therapy; Analysis of Covariance to test whether mean change in International Prostate Symptom Score from Baseline to 12 weeks differed among groups after controlling for baseline International Prostate Symptom Score and age. Last Observation Carried Forward was used to impute missing values; Test type: Superiority or Other; p = 0.2384, ANCOVA

ADVERSE EVENTS:
Time Frame: From Baseline through 12 Weeks
Arm/Group | Behavioral Treatment Alone | Drug Therapy Alone | Combined Behavioral + Drug Therapy
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/68 | 0/65
Serious Adverse Events (participants affected / at risk) | 1/71 | 2/68 | 1/65
Other Adverse Events (participants affected / at risk) | 0/71 | 0/68 | 0/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Treatment Alone (N=71) | Drug Therapy Alone (N=68) | Combined Behavioral + Drug Therapy (N=65)
Admittance to Hospital for Suicidal Thoughts (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Deemed unrelated to Behavioral Intervention
Taking too much study medication (General disorders) | 0 (0) | 1 (1) | 0 (0) — Subject within the Drug Only group misunderstood dosing regimen. No side effects observed, but reported to Internal Review Board (IRB) as Adverse Event
Admitted to Hospital for Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Subject within Drug Arm had a prior valve replacement 12 years prior to the study. Upon hospitalization, cardiology deemed a new valve was needed. It was deemed by the Data Safety Monitoring Board (DSMB), the Adverse Event was not related to study.
Admission to Hospital for Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Patient within the Combined Arm was admitted to hospital for observation due to shortness of breath. Patient was discharged, expressed desire to continue in the study. DSMB concluded adverse event was not associated with study or study drug.

LIMITATIONS AND CAVEATS:
No limitations or caveats for this trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No